CLINICAL TRIAL: NCT05249296
Title: The Impact of Green Spaces on the General Well-being and Stress of Students: an Intervention Study
Brief Title: The Impact of Green Spaces on the General Well-being and Stress of Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Michelle Plusquin, assistant professor, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Nature_Stress
Record Dates: First submitted 2020-04-02; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Stress; Neurocognition; Psychological; Cardiovascular
Keywords: Green space

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: intervention/control group (Experimental): Phase 1: Two weeks of green space intervention
  Phase 2: One week wash out period Resume daily activities
  Phase 3: Two weeks of 'daily activities' Regular, daily activities are resumed by the participants
  Phase 4: One week wash out period Resume daily activities
  Between each phase, detailed questionnaires, neurocognitive tests and cardiovascular measurements are taken from the participants.
  Interventions: Other: Nature based solution for stress reduction
- Group 2: control/intervention group (Experimental): Phase 1: Two weeks of 'daily activities' Regular, daily activities are resumed by the participants
  Phase 2: One week wash out period Resume daily activities
  Phase 3: Two weeks of green space intervention
  Phase 4: One week wash out period Resume daily activities
  Between each phase, detailed questionnaires, neurocognitive tests and cardiovascular measurements are taken from the participants.
  Interventions: Other: Nature based solution for stress reduction

INTERVENTIONS:
Other: Nature based solution for stress reduction — participation in nature activities: daily 30 min walking in nature

SUMMARY:
The number of students with psychological problems is on the rise, due to a combination of increasing performance pressure, high expectations, difficulties handling stress, social pressure, and studying. Spending time in a green space has been shown to have positive effects on the mental and general health. This project aims to alleviate the symptoms of mental fatigue and stress related disorders such as burn out in students by offering a nature-based activity.

Participants are asked to take a thirty-minute walk in a nature-based area for five consecutive days, followed by a control period (regular schedule of the participant) for five days, or vice versa. The investigators test stress-related parameters including concentration tests, cognitive tests, cortisol levels, and cardiovascular measurements.

DETAILED DESCRIPTION:
This project aims study the effectiveness of nature-based solutions on the prevention of stress-related symptoms due to high study pressure in students. A nature-based physical activity is recommended once a day to prevent stress build-up and positively influence the cardiovascular system. Participants are randomized into two groups: the first group of participants are asked to walk a nature-based route near the University campus for thirty minutes per day for two weeks (phase 1). After each activity-based phase, a washout period of one week is implemented to avoid carry-over of results (phase 2 and 4). In the third phase, the participants are asked to resume their daily activities for two weeks (control). The second group undergo the same phases but reversed: participants start with two weeks of their usual daily activities, followed by two weeks of nature-based activity. After each phase, the investigators measure neurocognition through neurocognitive tests, the emotional status through detailed questionnaires and assess stress levels through cardiovascular measurements, including salivary cortisol levels of saliva collected upon awakening, 30 min after waking and at 8 pm.

ELIGIBILITY:
Inclusion Criteria:

* Student of Hasselt university or university college PXL and dutch speaking

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
General health | 5 minutes
  An questionnaire is used to collect sociodemographic data and life-style factors, including movement data and health of the participant
Stress levels | 10 minutes
  Assessed via questionnaires (the burn out assessment tool (score 1-5) and general health questionnaire (score 0-12) and Five Item Well Being Index (score 0-100). Scores are used as continuous variables. Lower scores represent a lower risk of burn out, higher scores represent a higher risk of burnout. The score is constructed from questions concerning exhaustion, mental distance, emotional disorder(s), and cognitive disorder(s).
cortisol level (stress levels) | 5 minutes
  Assessed by salivary cortisol levels. Scale is µg/dl and used as a continuous variable.
visual memory | 5 minutes
  Computerized tests (eye-tracking test). The scale is pupil size, spontaneous blinking rate and eye movements and is used as a continuous variable.
selective attention | 5 minutes
  Computerized tests (stroop test). The scale is mean reaction time and is used as a continuous variable.
short-term memory | 10minutes
  Computerized tests (Digit Span Test). The scale is number of digits and is used as a continuous variable.
visual information processing speed | 5 minutes
  Computerized tests (Digit Symbol Test). The scale is number of digits and is used as a continuous variable.
visual information processing speed | 5 minutes
  Computerized tests (Pattern Comparison test). The scale is reaction time and is used as a continuous variable.
Heart rate variability | 30 minutes
  The heart rate is monitored throughout the entire baseline and follow-up visit through a small patch attached to the participant's skin. The results is used as a continuous variable in milliseconds (ms).
Blood pressure | 5 minutes
  Blood pressure is measured through an automated system. The results is used as a continuous variable in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Plusquin, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No
Data is pseudonymized. Data will then only be shared with the predoctoral researchers involved in this project, within our research group.